CLINICAL TRIAL: NCT06031337
Title: Salivary Expression of SOX7 in Oral Squamous Cell Carcinoma: Diagnostic Accuracy Study
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Salsabeel, Lecturer, Fayoum University
Other Study IDs: 1591985
Record Dates: First submitted 2023-09-02; First posted 2023-09-11 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Oral Cancer; Oral Squamous Cell Carcinoma
MeSH Terms: conditions — Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Oral Cancer Group: 23 patients with oral cancer
  Interventions: Diagnostic Test: ELISA
- Control Group: 23 age-and-sex-matched healthy individuals, as normal controls
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — quantitative determination of salivary SOX7 using an Enzyme Linked Immunosorbent assay (ELISA) kit based on the sandwich principle according to the manufacturer's protocol.

SUMMARY:
The study will include patients with oral cancer and healthy controls of both sexes. Subjects having any systemic diseases or other types of cancer will be excluded. All subjects will be selected from Oral Medicine Department, Faculty of Dentistry, Al Ahram Canadian University and Fayoum University. Informed consent will be obtained from all subjects enrolled in this study after explanation of the whole procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients with oral cancer

Exclusion Criteria:

* any systemic diseases or other types of cancer will be excluded

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 23 patients with oral cancer 23 healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2023-09-03 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
salivary expression of SOX7 | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
on request